CLINICAL TRIAL: NCT03760783
Title: The Effects of Microgravity on Human Sperm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Collaborators: Universitat Politècnica de Catalunya (Other); Dexeus Clinic Woman (Other)
Responsible Party: Principal Investigator, Montserrat Boada, Director of Reproductive Laboratory, Fundacion Dexeus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FSD-ATM-2018-03
Record Dates: First submitted 2018-11-15; First posted 2018-11-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Semen Quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of microgravity on human sperm (Other): Simulated microgravity flight
  Interventions: Other: Parabolic flight

INTERVENTIONS:
Other: Parabolic flight — Sperm analysis (total motility M/ml; grade a+b sperm M/ml, vitality, DNA Frag and apoptosis) will be measured on ground at 1g before the flight and after flight were sperm samples have been exposed to simulated microgravity

SUMMARY:
It has been described that microgravity affects cellular and molecular structures. Cell membrane, cytoskeleton, cytoplasm and nucleus have been found to be sensible to gravitational changes. Alterations in the male and female reproductive systems have also been reported in mouse and other animals. The effects of microgravity on human reproductive cells remain unknown.

The main objective of this experimental study is to investigate the effect of simulated microgravity in human male reproductive cells under in vitro conditions. Induced microgravity conditions will be obtained with a smaller single-engine aerobatic aircraft that can provide parabolic flights.

The main parameters to be analyzed are: sperm motility, vitality, DNA fragmentation and apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men)
* Who accepted to take part in the study
* Who gave their written informed consent

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Sperm motility | In earth gravity g=1(<4 hours before Parabolic flight) and after simulated microgravity exposure (<4 hours Post Parabolic Flight)
  The percentage of normal spermatozoa in terms of motility grades a,b,c according to WHO
Change Sperm Morphology | In earth gravity g=1(<4 hours before Parabolic flight) and after simulated microgravity exposure (<4 hours Post Parabolic Flight)
  The percentage of normal spermatozoa in terms of morphology is assessed by staining. The lower reference limit for normal forms is 4% (WHO 2010).
Change Sperm Vitality | In earth gravity g=1(<4 hours before Parabolic flight) and after simulated microgravity exposure (<4 hours Post Parabolic Flight)
  The percentage of live spermatozoa is assessed by identifying those with an intact cell membrane, from dye exclusion. The lower reference limit for vitality (membrane-intact spermatozoa) is 58% (WHO 2010).
Change in Sperm DNA Fragmentation | In earth gravity g=1(<4 hours before Parabolic flight) and after simulated microgravity exposure (<4 hours Post Parabolic Flight)
  Sperm DNA fragmentation is evaluated by Halosperm® kit, based on the SCD technique, patented by Halotech. This kit is based on a controlled DNA denaturation process to facilitate the subsequent removal of the proteins contained in each spermatozoon. In this way, normal spermatozoa create halos formed by loops of DNA at the head of the sperm, which are not present in those with damaged DNA.
  Thresholds for frequency of Sperm DNA Fragmentation (SDF) have been suggested by Dr. Evenson et al. (Evenson and Nixon, Reprod Biomed Online 12:466-472, 2006). The authors reported that couples with no known infertility problems were more likely to achieve a pregnancy/delivery if the DNA fragmentation index (DFI) was <30%.
Change Sperm APOPTOSIS (Annexin V ) | In earth gravity g=1(<4 hours before Parabolic flight) and after simulated microgravity exposure (<4 hours Post Parabolic Flight)
  Annexin V recognizes an antigen (externalized phosphatidylserine, EPS) in the plasma membrane of apoptotic cells. Apoptotic cell depletion begins with the magnetic labeling of apoptotic cells by the MACS® ART Annexin V Reagent. The labeled cells are then passed through a separation column located in a fixed magnetic field. Unwanted cells are selectively retained in the column. Living spermatozoa are not labeled by the reagent, so they pass through the column and are collected for later use.
  In our study, after collecting living spermatozoa we also collected the retained apoptotic spermatozoa for comparing the concentration (M/ml) of apoptotic vs no apoptotic cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Dexeus Departament d'Obstetrícia, Ginecologia i Reproducció, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boada M, Perez-Poch A, Ballester M, Garcia-Monclus S, Gonzalez DV, Garcia S, Barri PN, Veiga A. Microgravity effects on frozen human sperm samples. J Assist Reprod Genet. 2020 Sep;37(9):2249-2257. doi: 10.1007/s10815-020-01877-5. Epub 2020 Jul 18. PMID 32683528
- See also: Related Info — https://www.dexeus.com/